CLINICAL TRIAL: NCT03628612
Title: Long-term Follow-up of Patients Previously Treated With Autologous T Cells Genetically Modified With Viral Vectors
Brief Title: Long-term Follow-up of Patients Treated With Genetically Modified Autologous T Cells
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Autolus Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AUTO-LT1
Record Dates: First submitted 2018-07-07; First posted 2018-08-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Patients Followed for up to 15 Years Following Their First Dose of AUTO CAR T Cell Therapy; Multiple Myeloma; DLBCL; ALL, Adult and Pediatric; T Cell Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AUTO CAR T cell therapy (Experimental): Patients who received previous treatment with AUTO CAR T Cell Therapy
  Interventions: Biological: AUTO CAR T cell therapy

INTERVENTIONS:
Biological: AUTO CAR T cell therapy — No study drug is administered in this study. Patients previously treated with AUTO CAR T cell therapy will be monitored for safety following the first infusion.

SUMMARY:
Long-term follow-up of patients exposed to an AUTO CAR T cell therapy for up to 15 years following their first AUTO CAR T cell therapy infusion.

DETAILED DESCRIPTION:
The purpose of this study is to monitor all patients exposed to an AUTO CAR T cell therapy, for up to 15 years following their first AUTO CAR T cell therapy infusion to assess the risk of delayed treatment-related SAEs, adverse events of special interest (AESIs), monitor for emergence of replication competent retrovirus (RCR) or replication competent lentivirus (RCL), monitor for the emergence of a new malignancy associated with insertional mutagenesis (insertion site analysis), assess CAR transgene persistence and assess long-term efficacy. Monitoring of such long-term effects of AUTO CAR T cell therapy will help to further define the risk-benefit profile of these new CAR T cell therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have received an AUTO CAR T cell therapy on a clinical treatment study.
2. Patients must have provided informed consent for long-term follow-up study prior to participation.
3. Patients must be able to comply with the study requirements.

Exclusion Criteria:

1. There are no specific exclusion criteria for this study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-08-02 (Actual); Primary Completion 2043-07 (Estimated); Study Completion 2043-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events (SAE), new malignancies & adverse events of special interest (AESI) related to AUTO CAR T cell therapy | For up to 15 years
  Monitoring of all SAEs / AESIs, including any new malignancy or new diagnosis of neurologic disorders, or other hematologic disorder, related to AUTO CAR T cell therapy.
  Monitoring of all adverse events of special interest related to AUTO CAR T cell therapy infusion.

SECONDARY OUTCOMES:
Overall Survival following first AUTO CAR T cell therapy infusion. | Month 3, Month 6, Month 9, Month 12 during Year 1 following AUTO CAR T cell therapy infusion, then every 6 months up to Year 5, then yearly up to Year 15
  Overall Survival following first AUTO CAR T cell therapy infusion.
Duration of supportive care | Month 3, Month 6, Month 9, Month 12 during Year 1 following AUTO CAR T cell therapy infusion, then every 6 months up to Year 5, then yearly up to Year 15
  B-cell aplasia for patients treated with an AUTO CAR T cell therapy targeting a B-cell malignancy.
Duration of response | Month 3, Month 6, Month 9, Month 12 during Year 1 following AUTO CAR T cell therapy infusion, then every 6 months up to Year 5, then yearly up to Year 15
  Clinical efficacy of AUTO CAR T cell therapy in patients enrolled prior to disease progression.
Progression-free survival | Month 3, Month 6, Month 9, Month 12 during Year 1 following AUTO CAR T cell therapy infusion, then every 6 months up to Year 5, then yearly up to Year 15
  Progression free survival following first AUTO CAR T cell therapy infusion.
Proportion of patients with detectable replication-competent retrovirus (RCR) or lentivirus (RCL) from first AUTO CAR T cell therapy infusion | For up to 15 years
  Monitor for the absence of detectable RCR or RCL after the first AUTO CAR T cell therapy infusion
Proportion of patients with detectable vector copy number (VCN) in peripheral blood | Month 3, Month 6, Month 9, Month 12 during Year 1 following AUTO CAR T cell therapy infusion, then every 6 months up to Year 5, then yearly up to Year 15
  Blood sample collection for VCN measurement to detect persistence of CAR transgene(s)
Testing for Insertional mutagenesis in case of a new malignancy | For up to 15 years
  Insertional site analysis of samples to determine insertional mutagenesis as a potential cause / contributor in case of a new malignancy.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - University of Miami, Miami, Florida
  - Washington University in St. Louis, St Louis, Missouri
  - St David's South Austin Medical Center, Austin, Texas
- United Kingdom (5):
  - Queen Elizabeth University Hospital, Glasgow
  - University College London Hospitals NHS Foundation Trust, London
  - Manchester Royal Infirmary Hospital, Manchester
  - Royal Manchester Children's Hospital, Manchester
  - Freeman Hospital, The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No